CLINICAL TRIAL: NCT05531136
Title: Effect of a Foot Muscle Strengthening Program in Mobile Older Adults Adults
Acronym: STIFF3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Reaching end of funding
Sponsor: Lydia Willemse (Other)
Collaborators: Fontys University of Applied Sciences (Other); KU Leuven (Other); Tilburg University (Other)
Responsible Party: Sponsor-Investigator, Lydia Willemse, MSc., Fontys University of Applied Sciences
Organization: Fontys University of Applied Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STIFF 3
Record Dates: First submitted 2022-07-26; First posted 2022-09-07 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Fall Risk
Keywords: falling; foot exercises; older adults; mobility

STUDY DESIGN:
Intervention Model Description: The study design is an assessor-blinded RCT with two parallel groups. Participants are randomly assigned in a 1:1 ratio to either the intervention or the control group by the use of a computer-generated randomization list managed by an independent project administrator. Blocking, the size of the blocks undisclosed, is applied in order to ensure the balanced allocation at several time points in the trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Once a participant has accomplished the baseline measurements, the assessor requests group allocation. The project administrator then sends the allocation to the trainer, who assigns the participant to the allocated group. The nature of the intervention precludes blinding of the participants and the trainers, however staff members involved in the recruitment of participants and in the assessment of measurement variables remain blinded to the group allocation until the post-processing of data that involves any subjectivity has been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Foot strengthening training (Experimental): 12-week foot strengthening training in addition to an already joined functional exercise program. The foot strengthening training is supervised and progressing and consists of isolated and functional exercises. Participants keep a training diary.
  Interventions: Other: Foot strengthening training
- Control (No Intervention): The control group continues the functional exercise program as usual. The subjects in this group are asked to keep a diary in which the subjects weekly report other physical activities, fall incidents and mobility related discomfort. The trainer calls the participants in the control group every week to pay attention to these topics.

INTERVENTIONS:
Other: Foot strengthening training — a 12-weeks exercise program consisting of foot strengthening exercises prescribed for 5 daily sessions a week, of which 1 supervised, 20 minutes per session on top of the regular exercise therapy to prevent falling
  Arms: Foot strengthening training

SUMMARY:
Background of the study:

Falling is highly prevalent among older adults and has serious societal impact. Falls occur mainly during walking as a result of altered gait and/or the inability to maintain balance. The plantar intrinsic foot muscles (PIFM) have a role in these dynamic functions. When these muscles atrophy, as happens with advancing age, strengthening these muscles may be beneficial in order to improve or retain gait performance.

Objective of the study:

To investigate the effect of adding PIFM strengthening exercises to fall prevention programs compared to fall prevention programs alone on maximum gait speed in mobile older adults. The secondary objective is to also investigate the effect on: foot muscles' size, foot function during gait, balance during gait, discomfort during or after the training, self-reported mobility limitations, physical activity level, fall incidents during the intervention, fear of falling, foot plantar pressure during gait, static balance, toe flexor strength, physical functioning, foot morphology, foot posture.

Study design:

An investigator-blinded parallel randomized controlled trial (RCT), with a 12-week PIFM strengthening intervention period and pre- and post-intervention laboratory measurements.

Study population:

Older adults (>65 years) who are free of any known condition or disease that interferes with the execution of the exercise program.

Intervention:

Both the control and the intervention group continue with the regular exercise therapy to prevent falling. On top of this, the intervention group is delivered a 12-weeks exercise program consisting of foot strengthening exercises prescribed for 5 daily sessions a week, of which 1 supervised, 20 minutes per session.

Primary study parameters/outcome of the study:

The post-intervention difference between the intervention and control group in maximum gait speed.

Secondary study parameters/outcome of the study:

The post-intervention difference between the intervention and control group in foot muscles' size, foot function during gait, balance during gait, discomfort during or after the training, self-reported mobility limitations, physical activity level, fall incidents during the intervention, fear of falling, foot plantar pressure during gait, static balance, toe flexor strength, physical functioning, foot morphology, foot posture.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The burden for the participant consists mainly of 1) the time spent and effort put in engaging in the exercise therapy, 2) any discomfort (e.g., fatigue) or pain (e.g., cramp, muscle soreness) during or after the exercises, 3) the time that is spent on the measurement occasions (home visits: 1 x 1 hour (+ 1 x 30 minutes for the intervention group); laboratory: 2 x 3 hours), 4) the necessity of travelling to the motion analysis laboratory, 5) the inconvenience of wearing the activity monitor attached to the skin of the thigh for 7 days, and 6) questionnaires may unintentionally make the subject aware of declined health conditions.

ELIGIBILITY:
Inclusion Criteria:

* be 65 years of age or over;
* be able to ambulate 10 meter without using a walking aid;
* engage in a functional exercise program delivered to a group of older adults by an educated or certified physical therapist or trainer (e.g., fall preventive exercise program, senior fit programs);
* report to have 1) fear of falling OR 2) experienced a fall in the previous 12 months OR 3) difficulties with mobility, gait, or balance;
* be able to arrange their own transport to the movement analysis laboratory.

Exclusion Criteria::

* The respondent is a minor or legally incompetent adult;
* Self-reported presence of any disorder interfering with the execution of the exercises.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Maximum gait speed | 12 weeks
  The post-intervention difference between the intervention and control group in maximum gait speed.

SECONDARY OUTCOMES:
Foot muscles' morphology derived from ultrasound imaging | 12 weeks
Lower extremity biomechanics during gait assessed with 3D motion and ground reaction force capturing | 12 weeks
Spatiotemporal gait parameters assessed with 3D motion and ground reaction force capturing | 12 weeks
Balance during gait assessed with 3D motion and ground reaction force capturing | 12 weeks
Self-reported mobility limitations | 12 weeks
Weekly time spent in physical activities | 12 weeks
  in bouts of at least 10 minutes duration that is experienced by the participant at least as moderate intense (≥5 on a 10-point scale of how hard one feel he or she is exercising). From this it is deduced whether the participant meets the WHO recommendation on aerobic physical activity for health
Fall incidents during the intervention | 12 weeks
Fear of falling assessed by the (Falls Efficacy Scale-International) FES-I questionnaire | 12 weeks
Foot plantar pressure during gait assessed by a 2-meter pressure plate | 12 weeks
Static balance assessed by a force plate during single leg stance | 12 weeks
Isometric toe flexor strength assessed by a pressure plate during maximal toe press | 12 weeks
Physical functioning assessed by the Short Physical Performance Battery (SPPB) | 12 weeks
Foot arch characteristics assessed by a 3D foot scanner | 12 weeks
Health related quality of life assessed by SF-36 | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fontys Hogeschool, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Re-use of the data will be on request and on condition that all Principle Investigators agree and provided the requirements of the ethical committee are met

REFERENCES:
- [Derived] Willemse L, Wouters EJM, Pisters MF, Vanwanseele B. Effects of a 12-week intrinsic foot muscle strengthening training (STIFF) on gait in older adults: a parallel randomized controlled trial protocol. BMC Sports Sci Med Rehabil. 2024 Jul 20;16(1):158. doi: 10.1186/s13102-024-00944-z. PMID 39033125